CLINICAL TRIAL: NCT02715453
Title: Randomized Comparison Between a Strategy of Intervention in Frailty Versus the Usual Care in Frail Patients After an Acute Myocardial Infarction
Brief Title: Intervention in Frailty Versus Usual Care in Frail Patients After an Acute Myocardial Infarction
Acronym: FRAMIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan Sanchis, Prof, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/00837
Record Dates: First submitted 2016-03-04; First posted 2016-03-22 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Fragility
Keywords: Frailty; Acute myocardial infarction
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention on frailty (Experimental): Intervention on frailty in addition to the usual care by the cardiologist. A multidisciplinary team (physicians, nurses and physiotherapists and nutritionists) will carry out the intervention on frailty
  Interventions: Other: Intervention on frailty
- Control (No Intervention): Conventional strategy consisting only of the usual care by the cardiologist

INTERVENTIONS:
Other: Intervention on frailty — Multidisciplinary team (physicians, nurses, physiotherapists, and nutritionists):
  * Nutritional evaluation and intervention after randomization and regularly during follow-up
  * Physiotherapy sessions for 3 months after randomization and home exercise program for 1 year
  * Psychiatrist or psychologist assistance for 1 year after discharge
  Arms: Intervention on frailty

SUMMARY:
Frailty has been associated to a worse outcome in acute coronary syndromes, but the best management of frail patients after an acute coronary syndrome remains unknown. The aim was to investigate the benefit of an intervention on frailty in frail patients after an acute myocardial infarction.

Patients survivors after an acute myocardial infarction (with and without ST-segment elevation), older than 70 years and with pre-frailty (1-2 points) or frailty (≥3 points) according to the Fried's scale measured 24 hours before hospital discharge, will be included. The participants will be randomized to 2 strategies: a) intervention on frailty in addition to the usual care by the cardiologist, and b) conventional strategy consisting only of the usual care by the cardiologist. A multidisciplinary team (physicians, nurses and physiotherapists and nutritionists) will carry out the intervention on frailty The study contemplates a 2-year inclusion period and a 3rd year for the follow-up of the last included patient. The main outcome will be the frailty status (Fried's scale) at 3 months and 1 year. The secondary endpoint will be the clinical events, both cardiovascular and not cardiovascular events, including recurrent events (cumulative events analysis), for the total follow up (3 years in the case of the first included patient). The hypothesis is that an intervention on frailty will improve frailty status and the clinical outcomes in frail patients after an acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute myocardial infarction and survivors in the hospitalization phase
* Age =>70 years
* Prefrail or frail status (Fried scale =>1 points)

Exclusion Criteria:

* Cognitive impairment (Pfeiffer test)
* Severe concomitant disease that could hamper the participation in the study
* Patient refusal to participate

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01; Primary Completion 2019-08 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change on frailty status according to the Fried scale | 3 months and 1 year
  Points in the Fried scale

SECONDARY OUTCOMES:
Total cardiac (cardiac death, reinfarction, postdischarge revascularization, readmission for acute heart failure, readmission for other cardiac cause) and non-cardiac (all-cause mortality or readmission for non-cardiac cause) clinical events | Up to 3 years
  Number of participants with the events
All-cause mortality | Up to 3 years
  Number of participants dead
Ischemic events (reinfarction or postdischarge revascularization) | Up to 3 years
  Number of participants with reinfarction (readmission for chest pain with troponin elevation) or postdischarge revascularization (percutaneous coronary intervention or coronary surgery)
Readmission for acute heart failure | Up to 3 years
  Number of participants with readmission for acute heart failure
Readmission for non-cardiac causes | Up to 3 years
  Number of participants with readmission for non-cardiac cause
Change of Quality of life (EUROQOL) | 3 months and 1 year
  EUROQOL test
Change of Functional capacity (walk distance test) | 3 months and 1 year
  Distance walked during 6 minutes
Change of Nutritional status (Mini Nutritional Assessment) | 3 months and 1 year
  Mini Nutritional Assessment Test

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Sanchis, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanchis J, Nunez E, Ruiz V, Bonanad C, Fernandez J, Cauli O, Garcia-Blas S, Mainar L, Valero E, Rodriguez-Borja E, Chorro FJ, Hermenegildo C, Nunez J. Usefulness of Clinical Data and Biomarkers for the Identification of Frailty After Acute Coronary Syndromes. Can J Cardiol. 2015 Dec;31(12):1462-8. doi: 10.1016/j.cjca.2015.07.737. Epub 2015 Aug 21. PMID 26514748
- [Background] Sanchis J, Bonanad C, Ruiz V, Fernandez J, Garcia-Blas S, Mainar L, Ventura S, Rodriguez-Borja E, Chorro FJ, Hermenegildo C, Bertomeu-Gonzalez V, Nunez E, Nunez J. Frailty and other geriatric conditions for risk stratification of older patients with acute coronary syndrome. Am Heart J. 2014 Nov;168(5):784-91. doi: 10.1016/j.ahj.2014.07.022. Epub 2014 Jul 30. PMID 25440808
- [Derived] Sanchis J, Sastre C, Ruescas A, Ruiz V, Valero E, Bonanad C, Garcia-Blas S, Fernandez-Cisnal A, Gonzalez J, Minana G, Nunez J. Randomized Comparison of Exercise Intervention Versus Usual Care in Older Adult Patients with Frailty After Acute Myocardial Infarction. Am J Med. 2021 Mar;134(3):383-390.e2. doi: 10.1016/j.amjmed.2020.09.019. Epub 2020 Oct 24. PMID 33228950